CLINICAL TRIAL: NCT03303586
Title: Investigating the Effects of Wearing Compression Stockings to Improve Asthma Symptoms at Night
Brief Title: Effects of Compression Stockings in Asthma Symptoms at Night
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Azadeh Yadollahi, Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-5845-0
Record Dates: First submitted 2017-10-02; First posted 2017-10-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Asthma
Keywords: Asthma; Fluid Shift; Compression stockings; intrathoracic airway narrowing
MeSH Terms: conditions — Asthma | interventions — Stockings, Compression

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to wearing compression stockings for next two weeks or not wearing compression stockings for next two weeks, and crossed over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Asthma group (Active Comparator): Participants will be randomized to wear compression stockings or to control group for two weeks and cross over in the end of the period. When assigned to wear compression stockings, they will be instructed to put the stockings on as soon as they get up in the morning and to remove them just prior to bedtime for two weeks. If they have become loose, a new pair will be fitted. They will be given a diary to record the time they put on and remove the compression stockings each day. They will be telephoned after one week to check the fit of the compression stockings.
  Interventions: Other: Compression Stockings; Other: Control
- Healthy group (Active Comparator): Participants will be randomized to wear compression stockings or to control group for two weeks and cross over in the end of the period. When assigned to wear compression stockings, they will be instructed to put the stockings on as soon as they get up in the morning and to remove them just prior to bedtime for two weeks. If they have become loose, a new pair will be fitted. They will be given a diary to record the time they put on and remove the compression stockings each day. They will be telephoned after one week to check the fit of the compression stockings.
  Interventions: Other: Compression Stockings; Other: Control

INTERVENTIONS:
Other: Compression Stockings — We will use knee length, ready-made compression stockings at a pressure of 20-30mmHg at the ankle and if a good fit cannot be obtained, custom-made stockings will be ordered. Patients will be measured for compression stockings by a certified fitter.
Other: Control — Participants will not wearing compression stockings for two weeks.

SUMMARY:
Nocturnal worsening of asthma is common. It is characterized by overnight exacerbation of asthma symptoms such as shortness of breath, chest tightness, coughing, and wheezing, increased need of asthma medications and airway hyperresponsiveness, and decline in lung function (1). Nocturnal asthma has been attributed in part to circadian variations in lung function and airway inflammation. However, other factors including sleep, supine posture and lung volume may also contribute to nocturnal asthma. Current treatments often improve nighttime asthma symptoms. Nevertheless, nocturnal asthma is still common. Up to 2/3rd of asthma patients report nocturnal asthma symptoms, and many asthma related events occur at night, indicating poor asthma control. Results from an ongoing study suggest that in asthma while subjects were supine, fluid shifted out of the legs and accumulated in the thorax (rostral fluid shift) contributing to lower airway narrowing in asthma. A previou study has shown that wearing compression stockings during the day reduces fluid retention in the legs, reduces nocturnal rostral fluid shift out of the legs, and improves sleep apnea (2, 3). The aims of the proposed study is investigate whether off-the-shelf, below the knee compression stockings will attenuate nocturnal fluid shift and lower airway narrowing in asthma.

ELIGIBILITY:
Inclusion Criteria: non-smokers or former smokers (<10 pack/year)

Exclusion Criteria: uncontrolled hypertension

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Effect of wearing compression stockings on reducing rostral fluid shift during sleep and its effect in airway narrowing | After 2 weeks of the intervention
  Effect of wearing compression stockings or not on reducing fluid retention in the legs, reducing rostral fluid shift during sleep and improving nocturnal lower airway narrowing in asthma. After 2 weeks using or not compression stockings we will measure the overnight fluid volumes changes in leg, thorax and neck; changes in the respiratory impedance, pulmonary diffusion capacity and lung volume pre and post night of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Azadeh Yadollahi, Principal Investigator — Scientist
Locations (1):
- Toronto Rehabilitation Institute (TRI), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skloot GS. Nocturnal asthma: mechanisms and management. Mt Sinai J Med. 2002 May;69(3):140-7. PMID 12035073
- [Background] Redolfi S, Arnulf I, Pottier M, Lajou J, Koskas I, Bradley TD, Similowski T. Attenuation of obstructive sleep apnea by compression stockings in subjects with venous insufficiency. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1062-6. doi: 10.1164/rccm.201102-0350OC. PMID 21836140
- [Background] White LH, Lyons OD, Yadollahi A, Ryan CM, Bradley TD. Effect of below-the-knee compression stockings on severity of obstructive sleep apnea. Sleep Med. 2015 Feb;16(2):258-64. doi: 10.1016/j.sleep.2014.12.005. Epub 2014 Dec 18. PMID 25620198
- [Background] Theriault L, Hermus G, Goldfarb D, Stonebridge C, Bounajm F. Cost Risk Analysis for Chronic Lung Disease in Canada. The Conference Board of Canada, 2012.
- [Background] Braido F, Baiardini I, Ghiglione V, Fassio O, Bordo A, Cauglia S, Canonica GW. Sleep disturbances and asthma control: a real life study. Asian Pac J Allergy Immunol. 2009 Mar;27(1):27-33. PMID 19548627
- [Background] Turner-Warwick M. Epidemiology of nocturnal asthma. Am J Med. 1988 Jul 29;85(1B):6-8. doi: 10.1016/0002-9343(88)90231-8. PMID 3400687
- [Background] Robertson CF, Rubinfeld AR, Bowes G. Deaths from asthma in Victoria: a 12-month survey. Med J Aust. 1990 May 21;152(10):511-7. doi: 10.5694/j.1326-5377.1990.tb125350.x. PMID 2338923
- [Background] Yadollahi A, Singh B, Bradley TD. Investigating the Dynamics of Supine Fluid Redistribution Within Multiple Body Segments Between Men and Women. Ann Biomed Eng. 2015 Sep;43(9):2131-42. doi: 10.1007/s10439-015-1264-0. Epub 2015 Jan 30. PMID 25632892
- [Background] Thomas M, Kay S, Pike J, Williams A, Rosenzweig JR, Hillyer EV, Price D. The Asthma Control Test (ACT) as a predictor of GINA guideline-defined asthma control: analysis of a multinational cross-sectional survey. Prim Care Respir J. 2009 Mar;18(1):41-9. doi: 10.4104/pcrj.2009.00010. PMID 19240948
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Chung F, Abdullah HR, Liao P. STOP-Bang Questionnaire: A Practical Approach to Screen for Obstructive Sleep Apnea. Chest. 2016 Mar;149(3):631-8. doi: 10.1378/chest.15-0903. Epub 2016 Jan 12. PMID 26378880
- [Background] Netzer NC, Stoohs RA, Netzer CM, Clark K, Strohl KP. Using the Berlin Questionnaire to identify patients at risk for the sleep apnea syndrome. Ann Intern Med. 1999 Oct 5;131(7):485-91. doi: 10.7326/0003-4819-131-7-199910050-00002. PMID 10507956
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] Chen MJ, Fan X, Moe ST. Criterion-related validity of the Borg ratings of perceived exertion scale in healthy individuals: a meta-analysis. J Sports Sci. 2002 Nov;20(11):873-99. doi: 10.1080/026404102320761787. PMID 12430990
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Hlatky MA, Boineau RE, Higginbotham MB, Lee KL, Mark DB, Califf RM, Cobb FR, Pryor DB. A brief self-administered questionnaire to determine functional capacity (the Duke Activity Status Index). Am J Cardiol. 1989 Sep 15;64(10):651-4. doi: 10.1016/0002-9149(89)90496-7. PMID 2782256
- [Background] Zhang B, Lewis SM. A study of the reliability of clinical palpation of the spleen. Clin Lab Haematol. 1989;11(1):7-10. doi: 10.1111/j.1365-2257.1989.tb00168.x. PMID 2706905
- [Background] Cavalcanti JV, Lopes AJ, Jansen JM, Melo PL. Detection of changes in respiratory mechanics due to increasing degrees of airway obstruction in asthma by the forced oscillation technique. Respir Med. 2006 Dec;100(12):2207-19. doi: 10.1016/j.rmed.2006.03.009. Epub 2006 May 18. PMID 16713226
- [Background] Desjardin JA, Sutarik JM, Suh BY, Ballard RD. Influence of sleep on pulmonary capillary volume in normal and asthmatic subjects. Am J Respir Crit Care Med. 1995 Jul;152(1):193-8. doi: 10.1164/ajrccm.152.1.7599823.
- [Background] ROUGHTON FJ, FORSTER RE. Relative importance of diffusion and chemical reaction rates in determining rate of exchange of gases in the human lung, with special reference to true diffusing capacity of pulmonary membrane and volume of blood in the lung capillaries. J Appl Physiol. 1957 Sep;11(2):290-302. doi: 10.1152/jappl.1957.11.2.290. No abstract available. PMID 13475180
- [Background] Hsia CC. Recruitment of lung diffusing capacity: update of concept and application. Chest. 2002 Nov;122(5):1774-83. doi: 10.1378/chest.122.5.1774. PMID 12426283
- [Background] Stickland MK, Lindinger MI, Olfert IM, Heigenhauser GJ, Hopkins SR. Pulmonary gas exchange and acid-base balance during exercise. Compr Physiol. 2013 Apr;3(2):693-739. doi: 10.1002/cphy.c110048. PMID 23720327
- [Background] Huang YC, Helms MJ, MacIntyre NR. Normal values for single exhalation diffusing capacity and pulmonary capillary blood flow in sitting, supine positions, and during mild exercise. Chest. 1994 Feb;105(2):501-8. doi: 10.1378/chest.105.2.501. PMID 8306754
- [Background] Rosenberg E. The 1995 update of recommendations for a standard technique for measuring the single-breath carbon monoxide diffusing capacity (transfer factor). Am J Respir Crit Care Med. 1996 Jul;154(1):265-6. doi: 10.1164/ajrccm.154.1.8680694. No abstract available.
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Fredberg JJ, Wohl ME, Glass GM, Dorkin HL. Airway area by acoustic reflections measured at the mouth. J Appl Physiol Respir Environ Exerc Physiol. 1980 May;48(5):749-58. doi: 10.1152/jappl.1980.48.5.749. PMID 7451282
- [Background] Fabra-Campos H. [Ionomer as a substitute for lost dentin in conservative dentistry]. Rev Eur Odontoestomatol. 1990 Sep-Oct;2(5):335-44. Spanish. PMID 2094267
- [Background] Bhatawadekar SA, Inman MD, Fredberg JJ, Tarlo SM, Lyons OD, Keller G, Yadollahi A. Contribution of rostral fluid shift to intrathoracic airway narrowing in asthma. J Appl Physiol (1985). 2017 Apr 1;122(4):809-816. doi: 10.1152/japplphysiol.00969.2016. Epub 2017 Jan 12. PMID 28082337